CLINICAL TRIAL: NCT04259723
Title: Virtual Reality Assisted Conscious Sedation During Transcatheter Aortic Valve Implantation - a Randomized Pilot Study
Brief Title: Virtual Reality Assisted Conscious Sedation During TAVI
Acronym: TAVI_VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-007
Record Dates: First submitted 2020-01-29; First posted 2020-02-06 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Severe Aortic Valve Stenosis; Anxiety; Pain
Keywords: TAVI; VR; 3D glasses
MeSH Terms: conditions — Aortic Valve Stenosis; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: VR during TAVI
- Control (No Intervention)

INTERVENTIONS:
Other: VR during TAVI — Virtual Reality (VR) glasses
  Arms: Intervention

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is an established therapy for patients with severe aortic valve stenosis. Pain and anxiety are major contributors to procedural complications. Virtual Reality (VR) glasses have already been used successfully in different clinical settings to treat anxiety and delirium. The aim of this prospective, randomized investigation is to prove the feasibility and safety of VR interventions in patients undergoing conscious sedation during TAVI with local anesthesia only.

ELIGIBILITY:
Inclusion Criteria:

* Interventional transfemoral TAVI
* Informed consent
* Normal or corrected vision (through glasses)

Exclusion Criteria:

* Patients whose communication is limited due to a language barrier
* Patients who could not watch the 3D video due to uncorrectable vision
* all patients with transapical TAVI were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | at Baseline
  A visual analog scale will be used to determine the level of anxiety before and after the procedure. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points (0=no anxiety, 10=maximum anxiety/extremly anxious)
Change in anxiety | after 24 hours
  A visual analog scale will be used to determine the level of anxiety before and after the procedure. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points (0=no anxiety, 10=maximum anxiety/extremly anxious)

SECONDARY OUTCOMES:
Time of VR | at Baseline
  The time [min] of VR use will be recorded during the procedure
Evaluation of clinical frailty scale | at Baseline
  The Clinical Frailty Scale (CFS) is a simple model visually describing patients physical conditions with nine classes from very fit (class 1) to terminally ill (class 9).
Measurement of pain: visual analog scale | after 24 hours
  A visual analog scale will be used to determine the level of pain after the procedure. A visual analog scale will be used to determine the level of anxiety before and after the procedure. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points (0=no pain, 10=unbearable pain)
Length of stay at hospital | up to 5 days
  The length of stay at hospital will be recorded.
Occurence of vomitting | at Baseline, periprocedural and after 24 hours
  Patients will be asked during and after the procedure for safety problems with special regards to vomiting
Occurence of nausea | at Baseline, periprocedural and after 24 hours
  Patients will be asked during and after the procedure for safety problems with special regards to nausea
Rate of Intra-hospital mortality | up to 5 days
  The intra-hospital mortality will be assessed after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided